CLINICAL TRIAL: NCT07387952
Title: The Safety and Efficacy of Fecal Microbiota Transplantation Combined With Nutritional Intervention in the Treatment of Functional Constipation：a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-25PJ1600
Record Dates: First submitted 2025-08-06; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-08

CONDITIONS: Constipation - Functional; Fecal Microbiota Transplantation (FMT); Chronic Constipation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT with nutritional intervention group (Experimental): Fecal microbiota transplantation (FMT) is a method for treating imbalances in the intestinal microbiota, by extracting a portion of feces from a healthy individual that contains a diverse population of beneficial bacteria, processing it, and transplanting it into the digestive system of the recipient to restore a balanced intestinal microbiota. Nutritional intervention involves high dietary fiber preparation.
  Interventions: Procedure: FMT

INTERVENTIONS:
Procedure: FMT — In this group, colonoscopy is performed and a colostomy is placed in the ileocecal region. Bacterial infusion is performed for 3 days with 100ml graft per day. Within 30 minutes after receiving the microbiota transplantation, take the high dietary fiber preparation and dissolve it in water according to the instructions. Blood, stool, and colonoscopy-derived mucosal samples are collected before and after FMT and Researchers conduct follow-ups.
  Other Names: FMT with nutritional intervention

SUMMARY:
Chronic constipation is a common gastrointestinal disease with a global prevalence of about 15%, significantly affecting daily life and quality of life. Traditional treatments primarily rely on laxatives, which may lead to adverse effects with prolonged use, while surgical interventions have limited patient acceptance. Recent studies indicate that gut microbiota therapies-including probiotics, prebiotics, synbiotics, postbiotics, and fecal microbiota transplantation (FMT)-can effectively manage chronic constipation. This study aims to investigate the safety and efficacy of FMT combined with a prebiotic nutritional intervention (using a co-localization strategy) in the treatment of functional constipation. Additionally, the investigators will explore changes in fecal microbiota and metabolomic profiles following the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 70.
2. Diagnostic criteria: Functional constipation (FC) in accordance with Rome IV criteria, which should meet the following conditions:

   * Symptom requirements: The following at least 2 items should occur in ≥25% of bowel movements: a. Straining during defecation; b. Hard stool (Bristol Stool Classification score 1-2); c. Feeling of incomplete evacuation; d. Rectal obstruction sensation; e. Need for finger assistance during defecation; f. Spontaneous bowel movements <3 times per week.
   * It is rare to have loose stools without laxatives.
   * Exclusion of irritable bowel syndrome (IBS): IBS diagnosis criteria not meeting Rome IV.
   * Disease course requirements: Symptoms persist for at least 6 months and meet the above criteria within the last 3 months.
3. Traditional treatment methods (dietary intervention, at least two laxatives or probiotics) are ineffective.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Unable to take the intervention product or complete the examination as required.
3. Language expression disorder or mental illness.
4. Physical examination showed severe liver and kidney dysfunction.
5. Acute gastrointestinal disease within 4 weeks.
6. Constipation caused by surgery in the past 4 weeks.
7. History or abnormal examination: cancer, severe enteritis, intestinal obstruction, inflammatory bowel disease, hypothyroidism, mental illness, stroke, heart disease, cirrhosis, renal failure, hematopoietic system diseases, organic bowel disease suggested by colonoscopy or imaging.
8. Participation in other clinical trials within 3 months prior to enrollment.
9. Other health problems are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Defecation (Spontaneous Bowel Movements) | Baseline, Weeks 4, 8, 12, 18, and 24
  The number of Spontaneous Bowel Movements (SBM) per week recorded by the participant in a diary.
Stool Consistency Assessed by Bristol Stool Form Scale (BSFS) | Baseline, Weeks 4, 8, 12, 18, and 24
  Stool consistency is evaluated using the Bristol Stool Form Scale. The scale ranges from Type 1 (Separate hard lumps) to Type 7 (Liquid consistency). Type 1 and 2 indicate constipation, while Type 3 and 4 are considered normal. Higher scores indicate looser stool consistency.
Severity of Defecation Straining | Baseline, Weeks 4, 8, 12, 18, and 24
  Patient-reported assessment of the effort required to defecate. Participants rate their straining severity on a scale (e.g., from 0 to 3, where 0 represents no straining and 3 represents severe straining). Higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From baseline through Week 24
  Number of participants with adverse events. Assessment includes monitoring for specific gastrointestinal symptoms (e.g., aggravation of diarrhea, abdominal discomfort/bloating) and systemic infections (e.g., secondary intestinal infection, bacteremia). Safety is assessed via telephone and offline visits.
Change in Gut Microbiota Composition Assessed by Metagenomic Sequencing | Baseline, Weeks 2, 4, 8, 12, 18, and 24
  Fecal samples are collected to analyze the changes in the gut microbiota structure. Analysis includes the relative abundance of bacterial species and diversity indices (e.g., Shannon index) using Metastats analysis to compare pre- and post-treatment compositions.

CONTACTS AND LOCATIONS:
Overall Officials: Jingnan Li, MD, Ph.D, Study Chair — Peking Union Medical College Hospital, Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No